CLINICAL TRIAL: NCT05148689
Title: A Double-blind, Randomized, Placebo Controlled Study, Comparing Oxymetazoline 1% Cream TO RHOFADE in the Treatment of Moderate to Severe Persistent Facial Erythema Assocoated With Rosacea
Brief Title: A Study Comparing Oxymetazoline 1% Cream to RHOFADE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XMTC-1810
Record Dates: First submitted 2021-11-23; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- test product (Experimental): Oxymetazoline Cream, 1%
  Interventions: Drug: Oxymetazoline hydrochloride Cream, 1%
- reference (Active Comparator): Rhofade™ (oxymetazoline) cream, 1%
  Interventions: Drug: Rhofade™ (oxymetazoline) cream, 1%
- placebo (Placebo Comparator): Vehicle of Test product
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxymetazoline hydrochloride Cream, 1% — Cream
  Other Names: Oxymetazoline
  Arms: test product
Drug: Rhofade™ (oxymetazoline) cream, 1% — cream
  Arms: reference
Drug: Placebo — cream
  Arms: placebo

SUMMARY:
randomized, double-blind, placebo controlled

DETAILED DESCRIPTION:
Subjects in this randomized, double-blind, placebo controlled study will be randomly assigned to treatment sequences with the test product, reference product or placebo control.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant female aged ≥18 years with a clinical diagnosis of facial rosacea;
2. Provided IRB approved written informed consent;
3. A CEA score of ≥3 prior to study drug application
4. A PSA score of ≥3 prior to study drug application

Exclusion Criteria:

1. Female subjects who were pregnant, nursing, or had planned to become pregnant during study participation;
2. History of hypersensitivity to the study product;
3. Presence of ≥3 facial inflammatory lesions of rosacea;
4. Particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, and isolated pustulosis of the chin);
5. Raynaud's syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, cerebral or coronary insufficiency, renal or hepatic impairment, scleroderma, Sjögren's syndrome, or depression;
6. Excessive facial hair (e.g., beards, sideburns, moustaches, etc.) that could interfere with diagnosis or study assessments;
7. Presence of significant hypertension or circulatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
erythema response success | 21 day
  at least a 2-grade improvement in both CEA and PSA

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Walker, Study Chair — WayCro / Trial Clinsultants
Locations (1):
- WAYcro, Dallas, Texas, United States